CLINICAL TRIAL: NCT05630976
Title: A SINGLE ARM, PROSPECTIVE, MULTI-CENTER STUDY TO EVALUATE SAFETY AND EFFICACY OF ISAVUCONAZOLE FOR PRIMARY TREATMENT OF CHINESE PATIENTS WITH INVASIVE FUNGAL DISEASE (IFD) CAUSED BY ASPERGILLUS SPECIES OR OTHER FILAMENTOUS FUNGI
Brief Title: Cresemba® in Treating Chinese Patients With IFD Caused by Aspergillus Species or Other Filamentous Fungi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3791001; NCT05630976 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Invasive Fungal Disease
Keywords: Isavuconazole; Invasive Aspergillus; Invasive mold
MeSH Terms: conditions — Invasive Fungal Infections | interventions — isavuconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isavuconazole (Experimental): This is a single arm study, all enrolled participants will receive the study medication.
  Interventions: Drug: Isavuconazole

INTERVENTIONS:
Drug: Isavuconazole — This is a single arm study, all enrolled participants will receive the study intervention.
  Other Names: Cresemba®

SUMMARY:
This study is a post-approval commitment study, and is designed to further evaluate the safety and efficacy of isavuconazole in a relatively larger Chinese population who will receive isavuconazole treatment in a post-marketing setting.

This is a single arm, prospective, multi-center study. This study is seeking Chinese patients with proven, probable or possible Invasive Fungal Disease (IFD) caused by Aspergillus species or other filamentous fungi. All the participants will receive isavuconazole treatment. The longest treatment duration in this study is 84 days (up to 180 days for participants diagnosed with IM).

The primary objective is to characterize the safety and tolerability of isavuconazole through observing the treatment emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

* proven, probable, or possible IFD caused by Aspergillus species, Mucorales species or other filamentous fungi
* body weight >40 kg at screening

Exclusion Criteria:

* either chronic aspergillosis, aspergilloma, or ABPA
* Advanced HIV infection with CD4 count < 200 or acquired immunodeficiency syndrome-defining condition
* people who are unlikely to survive 5 days or participants on mechanical ventilation
* severe hepatic impairment (Child-Pugh Class C)
* familial short QT syndrome
* Concomitant use of efavirenz, ritonavir, etravirine, rifampicin/rifampin, rifabutin, nafcillin, ketoconazole, or St. John's Wort in the 5 days prior to first administration of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) by System Organ Class (SOC) | From Baseline to End of Study (EOS) and Prothrombin Time (PT)

SECONDARY OUTCOMES:
Percentage of all-cause mortality following primary treatment with isavuconazole. | Day 42 and Day 84
Crude rate of overall response at EOT | Day 42, and 84
  Responses based on the investigators' assessment at EOT
Crude rate of success of the clinical response at EOT | Day 42, and 84
  Responses based on the investigators' assessment at EOT
Crude rate of success of the mycological response at EOT | Day 42, and 84
  Responses based on the investigators' assessment at EOT
Crude rate success of the radiological responses at EOT | Day 42, and 84
  Responses based on the investigators' assessment at EOT
Number of Participants with TEAEs related to study intervention | Day 42, and 84
Number of Participants with TE Serious Adverse Event (SAEs) related to study intervention | Day 42, and 84
Number of Participants with TEAE leading to discontinuation of study intervention | Day 42, and 84
Number of Participants with TEAE leading to deaths | Day 42, and 84
Number of all deaths | Day 42, and 84
Number of Participants with Clinical Laboratory Abnormalities | Day 42, and 84
Number of Participants with Vital Signs Abnormalities | Day 42, and 84
Number of Participants with Abnormal Electrocardiogram (ECG) | Day 42, and 84
Number of Participants with Abnormal Eye Examination. | Day 42, and 84
Isavuconazole plasma concentration | Day 3, 7, 14, and EOT visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- China (14):
  - The First Affiliated Hospital of USTC, Anhui Province Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Henan provincial people's hospital, Zhengzhou, Henan
  - Liaocheng people's Hospital, Liaocheng, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Institute of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University, Hangzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Jiading Central Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3791001